CLINICAL TRIAL: NCT00127283
Title: Randomised, Double-Blind, Placebo Controlled, Multi-Centre, Parallel Groups Confirmatory Efficacy and Safety Trial of Activated Recombinant Factor VII (NovoSeven®/Niastase®) in Acute Intracerebral Haemorrhage
Brief Title: Recombinant Factor VIIa in Acute Intracerebral Haemorrhage
Acronym: FAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7ICH-1641; 2004-004202-24 (EudraCT Number)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eptacog alfa (activated)

SUMMARY:
This trial is conducted in Asia, Europe, Middle East, North America, Oceania, and South America.

The purpose of this study is to evaluate the treatment of Recombinant Factor VIIa (eptacog alfa (activated)) in patients with acute intracerebral bleeding. It is expected that more patients will recover without severe permanent disability after acute treatment with Recombinant Factor VIIa by reducing further intracerebral bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracranial hemorrhage (ICH) within 3 hours after first symptom

Exclusion Criteria:

* Patients with secondary ICH
* Pre-existing disability
* Haemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Reducing disability and improving clinical outcome | After 3 months

SECONDARY OUTCOMES:
Reducing mortality
Reducing hematoma growth

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (146):
- United States (68):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Fort Smith, Arkansas
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Oceanside, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Stanford, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Englewood, Colorado
  - Novo Nordisk Investigational Site, Hartford, Connecticut
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Maywood, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Fort Wayne, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Golden Valley, Minnesota
  - Novo Nordisk Investigational Site, Blackwater, Mississippi
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Lebanon, New Hampshire
  - Novo Nordisk Investigational Site, Cherry Hill, New Jersey
  - Novo Nordisk Investigational Site, Hackensack, New Jersey
  - Novo Nordisk Investigational Site, Ridgewood, New Jersey
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Stony Brook, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Durham, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Allentown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Hashville, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Burlington, Vermont
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Madison, Wisconsin
- Australia (4):
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Camperdown
  - Novo Nordisk Investigational Site, Gosford
  - Novo Nordisk Investigational Site, Heidelberg Heights
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
- Belgium (3):
  - Novo Nordisk Investigational Site, Antwerp
  - Novo Nordisk Investigational Site, Bruges
  - Novo Nordisk Investigational Site, Brussels
- Brazil (2):
  - Novo Nordisk Investigational Site, Sao Cristóvao
  - Novo Nordisk Investigational Site, Vila Clementino
- Canada (14):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Calgary
  - Novo Nordisk Investigational Site, Greenfield Park
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Mississauga
  - Novo Nordisk Investigational Site, Montreal
  - Novo Nordisk Investigational Site, Ottawa
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Saint John
  - Novo Nordisk Investigational Site, Saskatoon
  - Novo Nordisk Investigational Site, Thunder Bay
  - Novo Nordisk Investigational Site, Toronto
  - Novo Nordisk Investigational Site, Vancouver
- China (2):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Denmark (4):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Aarhus
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Glostrup Municipality
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Seinäjoki
  - Novo Nordisk Investigational Site, Turku
- France (3):
  - Novo Nordisk Investigational Site, Bordeaux
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Toulouse
- Germany (9):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, Minden
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Münster
- Novo Nordisk Investigational Site, Hong Kong, Hong Kong
- Israel (2):
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (4):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Pavia
  - Novo Nordisk Investigational Site, Perugia
  - Novo Nordisk Investigational Site, Roma
- Netherlands (5):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Heerlen
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Utrecht
- Norway (5):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Kristiansand
  - Novo Nordisk Investigational Site, Nordbyhagen
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Novo Nordisk Investigational Site, Singapore, Singapore
- Spain (4):
  - Novo Nordisk Investigational Site, Badalona
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Girona
  - Novo Nordisk Investigational Site, Madrid
- Sweden (4):
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Umeå
- Novo Nordisk Investigational Site, Lausanne, Switzerland
- Taiwan (2):
  - Novo Nordisk Investigational Site, Taipei
  - Novo Nordisk Investigational Site, Taoyuan District
- Novo Nordisk Investigational Site, Bangkok, Thailand

REFERENCES:
- [Result] Hsia CC, Chin-Yee IH, McAlister VC. Use of recombinant activated factor VII in patients without hemophilia: a meta-analysis of randomized control trials. Ann Surg. 2008 Jul;248(1):61-8. doi: 10.1097/SLA.0b013e318176c4ec. PMID 18580208
- [Result] Mayer SA, Brun NC, Begtrup K, Broderick J, Davis S, Diringer MN, Skolnick BE, Steiner T; FAST Trial Investigators. Efficacy and safety of recombinant activated factor VII for acute intracerebral hemorrhage. N Engl J Med. 2008 May 15;358(20):2127-37. doi: 10.1056/NEJMoa0707534. PMID 18480205
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com